CLINICAL TRIAL: NCT05113446
Title: A Prospective, Longitudinal Cohort Study of the Incidence of Dementia After the Onset of Delirium in Patients With Mild Cognitive Impairment: MDD Cohort (Mild Cognitive Impairment Delirium Dementia)
Brief Title: MDD(Mild Cognitive Impairment Delirium Dementia) Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Kyoung ja Moon, Assistant Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2019R1I1A3A0106056112
Record Dates: First submitted 2021-10-17; First posted 2021-11-09 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Delirium; Mild Cognitive Impairment; Dementia
Keywords: delirium; mild cognitive impairment; dementia
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MCI(Mild Cognitive Impairment) group: * Inclusion criteria : Patients 65 years of age or older who are admitted to a LTC(long-term care) facilities, Patients diagnosed with mild cognitive impairment by doctors, Patients with a score of 18 or more and 23 or less on the Mini-Mental State Examination
  * Exclusion criteria : Patients unable to measure the delirium assessment tool, The Short Confusion Assessment Methods (S-CAM) (Inouye, 2014) due to severe vision and hearing problems, Patients with serious psychiatric or neurological diagnosis,Patients who died or were transferred on the day of admission, Patients receiving emergency treatment at the time of the delirium assessment or unable to measure or intervene with S-CAM due to hospital circumstances
  Interventions: Diagnostic Test: Delirium assessment using S-CAM

INTERVENTIONS:
Diagnostic Test: Delirium assessment using S-CAM — Twice a day, the rounds of nurses in shifts, 8:00 am - 10:00 am, 4:00 pm - 6:00 pm Trained research assistants assessed delirium using S-CAM

SUMMARY:
* Identify the degree of delirium in subjects with mild cognitive impairment and find the risk factors of delirium. Mortality, hospital stay, and medical expenses are analyzed as clinical consequences related to delirium incidence.
* Dementia conversion rate and conversion period of subjects with mild cognitive impairment with delirium and it identifies the effect of delirium on dementia conversion.
* Develop an AI(Artificial intelligence) algorithm for predicting dementia transition in subjects with mild cognitive impairment based on the research results of the 1st, 2nd, and 3rd years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years of age or older who are admitted to a LTC
* Patients diagnosed with mild cognitive impairment by doctors
* Patients with a score of 18 or more and 23 or less on the Mini-Mental State Examination

Exclusion Criteria:

* Patients unable to measure the delirium assessment tool, The Short Confusion Assessment Methods (S-CAM) (Inouye, 2014) due to severe vision and hearing problems
* Patients with serious psychiatric or neurological diagnosis,Patients who expire or were transferred on the day of admission -
* Patients receiving emergency treatment at the time of the delirium assessment or unable to measure or intervene with S-CAM due to hospital circumstances

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to 3 long-term care (LTC) facilities
Sampling Method: Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Delirium incidence in participants with mild cognitive impairment | The number of subjects evaluated as positive in the delirium assessment using S-CAM for 30 days from the 1st day of study participation is statistically calculated.
  descriptive statistics
Dementia conversion rate and transition period in participants with mild cognitive impairment | The participant's dementia conversion is checked in units of 1 month, and the period until conversion to dementia is analyzed in units of 12 months for 36 months.
  descriptive statistics

SECONDARY OUTCOMES:
Risk factors affecting participants' delirium | On the first day of data collection, the characteristics of subjects are collected through medical records. After 12 months, the risk factors affecting the occurrence of delirium among the characteristics of the subject are analyzed.
  Logistic Regression
Mortality | It is statistically calculated in 30-day, 60-day, 12-month, 24-month, and 36-month increments.
  Kaplan-Meier survival, Cox proportional hazard regression, Logistic Regression
hospital length of stay | The period from hospitalization to discharge is calculated in days and analyzed in units of 12 months.
  Linear Regression
healthcare costs | From the healthcare costs consumed during the hospital length of stay, the direct healthcare costs used only for treatment are calculated in won units and analyzed in units of 12 months.
  Linear Regression

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Yangsan Seoul long-term care (LTC) facilities, Daegu, Gyeongsangnam-do
  - Gunsan Chamsarang long-term care (LTC) facilities, Daegu, Jeollabuk-do

REFERENCES:
- [Derived] Moon KJ, Park M. Protocol for a prospective, longitudinal cohort study on the incidence of dementia after the onset of delirium in patients with mild cognitive impairment: MDDCohort (Mild Cognitive Impairment Delirium Dementia). BMC Geriatr. 2024 Nov 7;24(1):922. doi: 10.1186/s12877-024-05480-6. PMID 39511473